CLINICAL TRIAL: NCT05839886
Title: The Adverse Event of Mitotane Therapy in Patients With Adrenocortical Carcinoma
Acronym: MEET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCEMD
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Adrenocortical Carcinoma
Keywords: Mitotane; Adverse effect
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This work will evaluate the adverse effects of mitotane treatment in patients treated for ACC with mitotane therapy. All of the individuals were treated at Ruijin Hospital between May 2023 and May 2024.

DETAILED DESCRIPTION:
Background: Adrenocortical Carcinoma (ACC) is a rare malignancy of the adrenal cortex. The annual incidence of ACC is thought to be between 0.5-2.0 cases per million. Adjunctive therapy with mitotane may be offered post- surgically to minimise risk of recurrence.

Aims: Evaluate the adverse effects of mitotane treatment in patients treated for ACC with mitotane therapy. All of the individuals were treated at Ruijin Hospital between May 2023 and May 2024.

Methods: Cortisol, ACTH, Gastrointestinal reactions and CNS Toxicity will be measured. SPSS v27 and GraphPad Prism v9.3.1 will be used for analysis and illustrations. Patients will be included, within ACC with mitotane. Data will be tested for normality, described as Mean± SD, compared using paired sample t-test with 5% p-value for significance and 95% confidence interval (CI).

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old and ≤ 75 years Diagnosis of Patients with adrenocortical cancer Gender: males and females Provide written informed consent Satisfactory compliance

Exclusion Criteria:

Patients with renal insufficiency (Cr>2 times the upper limit of normal). Patients with a history of liver cirrhosis. Patients who are currently using corticosteroids. Patients with cardiac insufficiency (NYHA cardiac function classification grade 3 and above or EF<50%).

Patients with stroke and acute myocardial infarction in the past 6 months. Patients during pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adrenocortical carcinoma treated with mitotane
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Documentation of adverse effects | from starting mitotane treatment until discontinuation of mitotane (since this is very variable from patient to patient no specific number of days or weeks can be entered (standard therapy would be about 2 years)
  Adverse effects will be documented using the NCI CTC AE v5

SECONDARY OUTCOMES:
Tumor treatment response | 2 years
  According to RECIST (version 1.1).